CLINICAL TRIAL: NCT00402441
Title: A One-Year, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Determine the Efficacy and Safety of 35-mg Risedronate Administered Once a Week in the Prevention of Osteoporosis in Postmenopausal Women
Brief Title: Risedronate in the Prevention of Osteoporosis in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HMR4003F/4001
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Risedronate (HMR4003)

SUMMARY:
Primary Objective:

* To demonstrate that risedronate 35-mg once weekly is more efficacious than placebo in increasing or maintaining bone mineral density (BMD) of the lumbar spine after 1 year of treatment in women who are non-osteoporotic and 0.5-5 years postmenopausal.

Secondary objectives:

* To demonstrate that risedronate 35-mg once weekly is more efficacious than placebo in increasing or maintaining total proximal femur, femoral neck, and trochanter BMD after 1 year of treatment in women who are 0.5-5 years postmenopausal
* To assess the general safety of 35-mg risedronate administered once weekly.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main Inclusion/Exclusion criteria are listed hereafter:

Inclusion criteria:

* Be postmenopausal for 0.5-5 years.Menopause is defined as 12 months without menses, based on medical history. Subjects who are post-menopausal secondary to bilateral oophorectomy must have serum FSH >40 mIU/mL and estradiol <20 pg/mL.
* Subjects with 3 contiguous lumbar spine vertebral bodies (L1-L4) without fracture or degenerative disease.
* Lumbar spine BMD mean value > 0.772g/cm2 (Hologic) or >0.880 g/cm2 (Lunar).

Exclusion criteria :

* Subjects with adequate lumbar spine BMD but osteoporotic by total proximal femur BMD (<0.637 g/cm2 [Hologic]) or <0.694 g/cm2 [Lunar]) as determined by dual-energy x-ray absorptiometry (DXA)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2002-09; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to Month12(endpoint) in lumbar spine BMD with imputation using LOCF principle.

SECONDARY OUTCOMES:
Percent change from baseline to Months 6 and 12 in lumbar spine BMD
and the percent change from baseline to Months 6, 12, and endpoint in total proximal femur, femoral neck, and trochanter BMD
Reported adverse events and changes in routine clinical laboratory tests, vital signs, and physical examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Matzkin, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States